CLINICAL TRIAL: NCT07119216
Title: The iPeer2Peer Support Mentorship Program for Young Adult Patients With Heart Disease: A Feasibility Study
Brief Title: The iPeer2Peer Mentorship Program for Young Adults With Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samantha Anthony (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor-Investigator, Samantha Anthony, Health Clinician Scientist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CTO5006; G-24-0036451 (Other Grant/Funding Number: Heart & Stroke Grant in Aid)
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Mentorship; Peer Support; Peer Support and Chronic Disease; Young Adults; Cardiomyopathies; Heart Transplant Recipient; Fontan Procedure
Keywords: heart failure; mentorship; peer support; young adult; heart disease
MeSH Terms: conditions — Heart Failure; Chronic Disease; Cardiomyopathies; Heart Diseases

STUDY DESIGN:
Intervention Model Description: A mixed methods pilot feasibility waitlist randomized controlled trial (RCT) design using central randomization with repeated measures, and following CONSORT guidelines, will be used to evaluate the iP2P program in young adult patients with heart disease. For clinical interventions, feasibility studies serve to identify potential refinements to the intervention, address uncertainties around the feasibility of intervention trial methods or test preliminary effects of the intervention. A waitlist pilot RCT allows for an effective comparison of the study intervention with a control group receiving standard of care while not disadvantaging the control group who will have the option of participating in the intervention following the completion of the trial.
Who Masked: Investigator
Masking Description: The randomization process will be blinded to the principal investigator and co-investigators to reduce the chance of experimenter bias. Mentees and mentors will be asked not to discuss their study involvement with others outside of the study team until study completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to their standard medical care, mentees in the experimental group will receive mentorship and support via the iP2P program. Trained mentors will provide information and support to mentee participants to encourage participation in self-management skill-building tailored to their needs. Each mentor will work with no more than two mentees at once for the study. Efforts will be made to pair mentors and mentees who share similar characteristics (e.g., similar disease severity, symptom profile, treatment regimen experiences, caregiver role, sex/gender, geographic area of residence). To ensure safety, a member of the research team will monitor all calls and messaging conversations as well as intervene in any potential safety concerns (e.g., discussion of suicidal ideation) or inappropriate behavior (e.g. bullying).
  Interventions: Behavioral: Peer Mentorship
- Waitlist control (No Intervention): The control group will receive standard care without the iP2P intervention. The control group will be offered the iP2P intervention after completion of all outcome measures for a period of 12 weeks with the same research team support.

INTERVENTIONS:
Behavioral: Peer Mentorship — The iPeer2Peer intervention is a peer support mentorship program that will provide modelling and reinforcement by pre-screened and trained peer mentors to the mentees. The mentorship program will encourage mentees to develop and engage in self-management and transition skills and support the participants; practice of these skills. The mentors will provide information and support to mentee participants via 5-10 calls (using WhatsApp) of 20-30 minute durations and text messaging (using WhatsApp) for 12 weeks to encourage participation in self-management skill building tailored to their needs.
  Other Names: Peer mentoring; Peer support
  Arms: Intervention group

SUMMARY:
Young adults with heart failure, including those who have undergone a heart transplant, experience considerable psychosocial stressors associated with living with a chronic illness, including heightened levels of anxiety and depression, and poor health-related quality of life compared to 'healthy' peers. Psychosocial challenges during young adulthood are especially concerning as this life stage represents a unique transitional period for fostering self-identity, friendships, mastery, and decision-making competencies. As young people with heart failure transition into adult healthcare systems, they take on greater personal responsibility due to their increasing independence and involvement in care decisions, and require more support and resources to live longer, healthier lives. Peer support provided by a person with a similar experience has been found to improve disease self-management and psychosocial health outcomes in pediatric healthcare.

An established, online mentorship program, iPeer2Peer (iP2P), will be employed through a pilot feasibility waitlist randomized controlled trial with repeated measures across five sites. Sixty mentees will be recruited and randomized into intervention and control groups. Thirty mentees in the intervention group will be matched 1:1 with 20 trained mentors. These pairings will connect over 12 weeks through video calls and text messaging to provide peer support to improve self-management and psychosocial health outcomes.

DETAILED DESCRIPTION:
Primary Objective: to evaluate the feasibility of the iP2P program in terms of participant: (a) recruitment and withdrawal rates, (b) adherence with the program, (c) perceptions regarding the acceptability and level of engagement in the iP2P program, and (d) perceptions of barriers and enablers of the iP2P program.

Secondary Objective: to explore the iP2P program's impact on preliminary psychosocial outcomes in:

i.Mentees- (a) disease self-management, (b) perceived social support, (c) emotional distress, (d) resiliency and (e) hope; ii.Mentors- (a) perceived social role satisfaction, (b) emotional distress, and (c) hope.

A waitlist pilot RCT allows for an effective comparison of the study intervention with a control group receiving standard of care while not disadvantaging the control group who will have the option of participating in the intervention following the completion of the trial.

Up to 80 participants will be enrolled in this study at five sites: Mazankowski Alberta Heart Institute (Edmonton), St. Boniface Hospital (Winnipeg), Toronto General Hospital (Toronto), the University of British Columbia Division of Cardiology - Vancouver General Hospital and St Paul's Hospital (Vancouver).

We expect 20 adult mentors and 60 young adult mentees will be enrolled across these sites, with 4-6 mentors and about 10-15 mentees per site. The mentees will be randomized to the experimental (iP2P program; n=30) or control (waitlist; n=30) group. Mentees assigned to the waitlist will receive the iP2P program once all outcome measures are complete.

All mentees will be asked to participate in semi-structured individual interviews at baseline (ME T1) and and all mentees in the intervention group will be asked to participate in semi-structured interviews at 12 weeks - immediately post-intervention (ME T2). Interviews will be conducted by an interviewer trained in qualitative methods by telephone, in-person or virtually via the PHIPA-compliant version of Zoom or Microsoft Teams (depending on participants' preference), at a time that is convenient for the participant. Interviews will be guided by a semi-structured interview guide. ME T1 interviews will aim to assess motivations for participation, hopes and expectations, and preferences around mentor characteristics; and ME T2 interviews will aim to assess the primary outcomes evaluating feasibility.

All mentors will be asked to participate in a focus group/semi-structured interview prior to mentor training (MR T1) and study end (MR T2). MR T1 focus groups/interviews will aim to assess motivations for participation and hopes and expectations, and MR T2 focus groups/interviews will aim to assess the primary outcomes evaluating feasibility. Focus groups/interviews will be conducted by an interviewer trained in qualitative methods. Focus groups/interviews will be conducted on a mutually agreed upon date and over the internet via a web-based video communication program (e.g., PHIPA-compliant version of Zoom or Microsoft Teams).

The semi-structured individual interviews and focus groups will be audiotaped, transcribed and analyzed using qualitative descriptive approach using thematic and content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Peer Mentor inclusion criteria: (a) heart disease patients, (b) at least three months post-diagnosis, (c) between the ages of 26-35 years old, (d) nominated by a member of their healthcare team as a good candidate to act in the mentor role based on maturity and emotional stability (e.g., good communication skills, positive adaptation and adjustment, strong support network), (e) willingness to commit to virtual peer mentor training, (f) able to speak and read English, and (g) access to a device (e.g., smart phone, tablet, computer) capable of using free WhatsApp software.
* Peer Mentee inclusion criteria: (a) heart disease patients, (b) between the ages of 18-25 years old, (c) able to speak and read English, and (d) access to a device (e.g., smart phone, tablet, computer) capable of using free WhatsApp software.

Heart disease patients include:

* Patients with any past or present heart failure
* Patients with cardiomyopathy seen at least 2 times a year
* Patients who have undergone a Fontan procedure
* Patients who have undergone a heart transplant

Exclusion Criteria:

* Mentor and mentee exclusion criteria include: (a) Significant cognitive impairments as assessed by a qualified healthcare provider (HCP), (b) have a diagnosis of an active psychological disorder (e.g.: Major Depressive Disorder, etc.; determined through chart review by a qualified HCP) likely to influence assessment of health-related quality of life and/or interfere with their ability to manage their heart disease care regimen, and (c) are participating in other peer support or self-management interventions.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment and withdrawal rates | Baseline to study completion
  (a) Recruitment rates (more than 70%) and withdrawal rates (less than 15%) as calculated using data recorded in participant recruitment log.
Level of engagement | 12 weeks
  Measured via semi-structured interviews or focus groups.
Adherence | 12 weeks
  More than 80% rate of completion of at least five audio or video calls over 12 weeks and 100% rate of completion of all online outcome measures as calculated using data recorded in participant program tracking log.
Acceptability | 12 weeks
  When the innovation is agreeable, palatable or satisfactory. Measured via focus groups or semi-structued interviews.
Barriers and enablers | 12 weeks
  Measured via semi-structued interviews or focus groups.

SECONDARY OUTCOMES:
Perceived social role satisfaction (Mentors) | Baseline to study completion, an average of 1 year
  Measured by the PROMIS Satisfaction with Social Roles and Activities
Emotional distress (Mentors) | Baseline to study completion, an average of 1 year
  Measured by the General Anxiety Disorder-7 and the Patient Health Questionnaire Depression Scale
Hope (Mentors) | Baseline to study completion, an average of 1 year
  Measured by the Adult Hope Scale
Disease self-management (Mentees) | Baseline to 12 weeks post-program completion and 24 weeks post-program completion
  Measured by the Partners in Health Scale
Percevied social support (Mentees) | Baseline to 12 weeks post-program completion and 24 weeks post-program completion
  Measured by the Multidimensional Scale of Perceived Social Support
Emotional distress (Mentees) | Baseline to 12 weeks post-program completion and 24 weeks post-program completion
  Measured by the General Anxiety Disorder-7 and the Patient Health Questionnaire Depression Scale
Resiliency (Mentees) | Baseline to 12 weeks post-program completion and 24 weeks post-program completion
  Measured by the Brief Resilience Scale
Hope (Mentees) | Baseline to 12 weeks post-program completion and 24 weeks post-program completion
  Measured by the Adult Hope Scale

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No